CLINICAL TRIAL: NCT05882526
Title: Comparative Evalutaion of the Efficiency of Maxillary Canine Retraction Using Orthodontic Elastomeric Chain Versus Burstone T-loop.A Clinical Study
Brief Title: Compartive Evalution of the Efficiency of Maxillary Canine Retraction Using Power Chain Versus Burstone T-loop
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelaziz Abdelaziz younes, investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: canine retraction in tooth
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Class I Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Intervention Model Description: Evaluation of T loop for orthodontic maxillary canine retraction Evaluation of POWER CHAIN for orthodontic maxillary canine retraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluation of elastomeric power chain for orthodontic maxillary canine retraction (Active Comparator): 20 Orthodontic patient treated by for elastomeric power chain canine retraction split mouth.
  Interventions: Device: BURSTONE T-LOOP
- Evaluation of T loop for orthodontic maxillary canine retraction (Active Comparator): 20 Orthodontic patient treated by T loop for canine retraction split mouth
  Interventions: Device: BURSTONE T-LOOP

INTERVENTIONS:
Device: BURSTONE T-LOOP — Split mouth study one side using elastomeric power chain and other side using T loops
  Other Names: elastomeric power chain

SUMMARY:
evaluate and compare the efficiency between elastomeric chains and burston T-loop retractors in terms of rate of maxillary canine retraction and canine movements

DETAILED DESCRIPTION:
The purpose of orthodontic treatment is to move teeth as efficiently as possible with minimal adverse effects on teeth and supporting tissue. Numerous methods of canine retraction are currently in common use. Force can be applied through the elastics, closed coil springs, wire loops of numerous designs, and a number of headgear types currently available.

The principles for retraction currently used in preadjusted edgewise mechanics can be described as either:(a) a frictional system in which the canine is expected to slide distally along a continuous archwire, (b) frictionless mechanics in which loops (springs) are incorporated in a continuous or a segmental archwire to retract teeth. The sliding mechanism in any application other than simple tipping movement has two disadvantages: (i) friction (ii)force magnitudes cannot be easily determined since the amount of friction is relatively unknown and unpredictable.1 Space closure in orthodontics is the second stage incomprehensive fixed appliance treatment and can be accomplished by either sliding mechanics or loop mechanics. Nickel-titanium closed-coil springs and elastomeric power chains (PC) are the most common force delivery systems used in space closure

In vitro studies of the properties of PC showed that they lose force much more rapidly than springs over time.2-3In addition, environmental factors and temperature have greater effects on the properties of PC than on CS.4 Arch-length-to-tooth-mass discrepancy patients require extraction of teeth and closure of those spaces to correct their malocclusion. There are different mechanical methods used in orthodontic practice to move teeth, such as using various types of elastic materials and coil springs5During the past few years, elastomeric power chains (EPCs) have been used in preference to other retraction orthodontic materials because of their elastic properties, ease of application and requiring no patient co-operation, low cost, being relatively hygienic, and their irritation-free nature due to their smooth surface6 The proper position of canines shares a very important role in oral function and esthetics. Their unique position makes their orthodontic movement of great clinical importance, especially in premolar extraction cases. Segmented arch technique is a modified edgewise orthodontic procedure developed by Burstone7 in 1962 which consists of multiple wires found in different portions of arch. The force systems are relatively constant and with long ranges of activation and optimum force levels their resulting movement is predictable, as stated by Burstone, Baldwin, Lawless.8 Later in 1966, Burstone CJ9 stated that moment-to-force ratio, magnitude of force and the constancy of force determine the success of an appliance. The segmented arch technique has many advantages like better control over the forces, more efficient tooth movement over long distances with light constant forces, as stated by Burstone, Koenig (1976).10 In 1980, Burstone and Goldberg11 introduced beta titanium molybdenum alloy (TMA) wire (11%molybdenum, 6% zirconium and 6% beta titanium alloy) which showed twice the amount of deflection and delivered half the amount of force as compared to stainless steel wires. Burstone, van Steenbergen, Hanley12 in 1995 mentioned that T-loops had three important characteristics, i.e."α" , i.e. anterior moment or β, i.e. posterior moment and a horizontal moment.

Viecilli (2006)13 stated that the effects of steps, angles and vertical forces could be combined to produce an ideal T-loop design. According to Proffit (2007),14 segmented retraction of canines with frictionless springs reduces the strain on posterior teeth. The T-loop design generally provides a constant moment:force (M:F) ratio, a light and constant force throughout the entire activation range of a closing loop, and a constant low load-deflection rate15

Canine retraction and space closure is considered the most time-consuming phase in orthodontic treatment.16 Acceleration of this step would reduce overall treatment time, improve patient cooperation, and decrease possible negative side effects.17,18 Manipulation of tooth biomechanics16-19and tissue reaction20 have been widely attempted to reduce treatment duration. Additionally, the rate and safety of different canine retraction methods20 and different force Various techniques for canine retraction have been introduced including Nickel Titanium closing coil, Elastomeric chains, and lace backs. On the other hand, frictionless mechanics imply the use of the sectional method as the use of Burstone's T - loop, Rickett's spring, or Gjessing's spring Researchers were interested in investigating the effect of different force levels on the rate of canine retraction using sectional springs. And many authors have described various designs of canine retraction springs, their suitability and efficiency 21,22

ELIGIBILITY:
Inclusion Criteria:

- Class I or bimaxillary protursion , orthodontic patients, with moderate to severe crowding who are indicated for maxillary first premolar extraction. 2- All permanent teeth are erupted (3rd molars are not included). 3- Good oral and general health. 4- No previous orthodontic treatment.

Exclusion Criteria:

- Orthodontic cases that could be treated with no indication for extraction therapy.

2- Orthodontic cases that are indicate for the extraction of any tooth other than maxillary first premolars. 3- Patients with systemic diseases that might interfere with the of orthodontic tooth movement.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
rate of canine retraction | FOUR months
  distance which canine move pre and post retraction
Canine rotation | 4 MONTH
  angulation of canine
canine tipping | 4 month
  canine movement in mesial and dISTAL

CONTACTS AND LOCATIONS:
Overall Officials: AHMED MAHER FOUDA, Study Chair — Mansoura University; nehal fouad elbelasy, Study Director — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barsoum HA, ElSayed HS, El Sharaby FA, Palomo JM, Mostafa YA. Comprehensive comparison of canine retraction using NiTi closed coil springs vs elastomeric chains. Angle Orthod. 2021 Jul 1;91(4):441-448. doi: 10.2319/110620-916.1. PMID 34181721
- [Result] Davis S, Sundareswaran S, James J. Comparative evaluation of the efficiency of canine retraction using modified Marcotte and T-loop retraction springs - A split-mouth, randomized clinical trial. J Orthod Sci. 2019 May 23;8:9. doi: 10.4103/jos.JOS_101_18. eCollection 2019. PMID 31161132